CLINICAL TRIAL: NCT02045550
Title: Tolerance and Effect of a Prophylactical Treatment With a Cough Medicine Con-taining Ivy Leaves Dry Extract in Children With Recurrent Wheezy Bronchitis
Brief Title: Tolerance and Effect of a Prophylactical Treatment With Ivy Leaves Dry Extract in Recurrent Wheezy Bronchitis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HeHe02
Record Dates: First submitted 2014-01-13; First posted 2014-01-27 (Estimated); Last update posted 2014-01-27 (Estimated); Status verified 2014-01

CONDITIONS: Acute Wheezy Bronchitis; Recurrent Bronchitis
MeSH Terms: conditions — Bronchitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo Syrup (Placebo Comparator): Placebo Syrup 2.5 ml twice daily for 4 weeks
- Prospan Syrup (Active Comparator): Prospan Syrup 2.5 ml twice daily for 4 weeks
  Interventions: Drug: Prospan Syrup

INTERVENTIONS:
Drug: Prospan Syrup — 2.5 ml twice daily for 4 weeks
  Arms: Prospan Syrup

SUMMARY:
To evaluate the effect of a prophylactical therapy with a cough medicine containing ivy leaves dry extract on the frequency of recurrent wheezy bronchitis in toddlers, on the duration of the bronchitis episodes, on the severity and the additional drug demand. A prolonged asymptomatic episode between each wheezy bronchitis due to the therapy is assumed.

ELIGIBILITY:
Inclusion Criteria:

1. Medical diagnosis of ≥3 episodes of wheezy bronchitis within the pre-vious 12 months
2. Children aged from 1 to 3 years (girls and boys)
3. Signed Informed Consent of the legal guardians to participate in the trial after written and verbal briefing by the Investigator
4. No allergic sensitization
5. Allowance to contact the familys pediatrician for medical history of wheezy bronchitis episodes

Exclusion Criteria:

1. Anamnestically known intolerance/allergy to one of the drugs applied or to their ingredients or to drugs of similar chemical structure
2. Participation of the patient in another clinical trial within the last four weeks before enrollment in this trial
3. Evidence suggesting that the patient or their legal representative is not likely to follow the trial protocol (e.g. lacking compliance)
4. Inability to document the symptoms in a symptom log book or ques-tionnaire; inability to take the trial medication properly
5. Any regular therapy except Vitamin D or Fluoride
6. Chronic illnesses of different aetiology
7. Premature birth or diagnosis of bronchopulmonary dysplasia
8. Gastro-oesophageal reflux
9. Hereditary fructose intolerance

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
the time to event (next bronchitis episode) rate during and after treatment period | three months

SECONDARY OUTCOMES:
days and percentage of days without bronchitis during and after treatment period | 3 months
days and percentage of days without bronchitis during treatment period | three months

CONTACTS AND LOCATIONS:
Overall Officials: Christian Vogelberg, MD PhD, Principal Investigator — Technische Universität Dresden
Locations (1):
- Universitätsklinikum Carl Gustav Carus, Klinik und Poliklinik für Kinder- und Jugendmedizin, Dresden, Saxony, Germany